CLINICAL TRIAL: NCT04868266
Title: A Randomized Controlled Trial of the Effect of Capnography for Preventing Hypoxia in Minimally Sedated Pediatric Patients
Brief Title: End Tidal Carbon Dioxide in Minimal Sedation
Acronym: ETCO2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D-2103-187-1208
Record Dates: First submitted 2021-04-25; First posted 2021-04-30 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Complication of Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- end tidal carbon dioxide monitoring (Experimental)
  Interventions: Other: end tidal carbon dioxide monitoring
- Oxygen saturation monitoring (No Intervention)

INTERVENTIONS:
Other: end tidal carbon dioxide monitoring — We will monitor end tidal carbon dioxide with capnography during minimal sedation
  Arms: end tidal carbon dioxide monitoring

SUMMARY:
This randomized controlled study investigated the effect of end-tidal carbon dioxide monitoring in pediatric patients undergoing minimal sedation.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing minimal sedation for procedure.

Exclusion Criteria:

* none

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 214 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of oxygen desaturation | from immediately after sedation to end of procedure, up to 2 hours
  oxygen saturation lower than 95%

SECONDARY OUTCOMES:
number of Staff intervetions | from immediately after sedation to end of procedure, up to 2 hours
  tactile stimulation, jaw thrust or head tilt, suction, oral or nasopharyngeal airway insertion, oxygen supply, laryngeal mask airway insertion, bag-valve mask ventilation, endotracheal intubation
Severe oxygen desaturation | from immediately after sedation to end of procedure, up to 2 hours
  oxygen saturation lower than 85%, 90%
Lowest oxygen saturation | from immediately after sedation to end of procedure, up to 2 hours
  value of oxygen saturation
Episode of apnea | from immediately after sedation to end of procedure, up to 2 hours
  capnography flat line more than 5 seconds
sedation level | from immediately after sedation to end of procedure, up to 2 hours
  6-point pediatric sedation state scale
inappropriate monitoring | from immediately after sedation to end of procedure, up to 2 hours
  the duration of inappropriate capnography monitoring
Airway obstruction | from immediately after sedation to end of procedure, up to 2 hours
  stridor, retraction
Integrated pulmonary index | from immediately after sedation to end of procedure, up to 2 hours
  calculated parameter
success of procedure | from immediately after sedation to end of procedure, up to 2 hours
  success or fail of sedation or procedure
Hemodynamic instability | from immediately after sedation to end of procedure, up to 2 hours
  heart rate and blood pressure change more than 20%
Medication | from immediately after sedation to end of procedure, up to 2 hours
  type and dosage of sedatives

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

REFERENCES:
- [Derived] Kim EH, Park JB, Ji SH, Jang YE, Lee JH, Kim HS, Kim JT. Using capnography in children to prevent oxygen desaturation during procedural sedation: A randomised trial. Eur J Anaesthesiol. 2025 Nov 1;42(11):1034-1041. doi: 10.1097/EJA.0000000000002250. Epub 2025 Aug 11. PMID 40810300